CLINICAL TRIAL: NCT03188120
Title: Specific Use-Result Surveillance of Spiriva Respimat in Asthmatics (Patients With Mild and Moderate Persistent Asthma)
Brief Title: Specific Use-Result of Spiriva Respimat® in Asthmatics
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0205-0536
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spiriva Respimat group
  Interventions: Drug: Spiriva Respimat

INTERVENTIONS:
Drug: Spiriva Respimat — Drug
  Other Names: FORVENT, SPIRIVA, SRIVASSO

SUMMARY:
The study objective is to investigate the safety and effectiveness of Spiriva Respimat in patients with mild to moderate persistent asthma under real-world use

DETAILED DESCRIPTION:
The study is Post-Marketing Surveillance on the Long-Term Use of Spiriva Respimat in Japanese patients with mild to moderate persistent asthma. The patient population who receive Spiriva Respimat and the safety profile is not expected to change. This study can investigate the safety and effectiveness of Spiriva Respimat in patients with mild to moderate persistent asthma under real-world use

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild to moderate persistent bronchial asthma
* Patient aged ≥ 15 years
* Patients who are naive to Spiriva Respimat and receive Spiriva Respimat for the first time for treatment of bronchial asthma on top of at least ICS treatment.

Exclusion Criteria:

* Patients who have a contraindication to Spiriva Respimat defined in the package insert for Spiriva Respimat
* Patients who have been enrolled in this study before.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with mild to moderate persistent bronchial asthma
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yukako Ogi, Study Chair — zzCDMJP_PV_PMS@boehringer-ingelheim.com
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, observational study to collect new real world data (i.e., data under routine medical practice) on safety and effectiveness of Spiriva Respimat treatment in patients.
Pre-assignment Details: All participants were screened for eligibility to participate in trial. They attended specialist sites to ensure that they (the participants) met all implemented inclusion/exclusion criteria. Participants were not to be entered to trial if any of the specific entry criteria was violated.
Groups:
- Spiriva Respimat Group: Patients with mild to moderate persistent asthma treated with Spiriva® 1.25 microgram (μg) Respimat® 60 puffs and Spiriva® 2.5 μg Respimat® 60 puffs (hereinafter, Spiriva Respimat). Daily dose was inhalation of the spray of two puffs of Spiriva 2.5 μg Respimat (5 μg of tiotropium) and the spray of two puffs of Spiriva 1.25 μg Respimat (2.5 μg of tiotropium) in this non-interventional, observational study to collect new real world data (i.e., data under routine medical practice)
Period: Overall Study
Arm/Group | Spiriva Respimat Group
Started (Case Report Form collected (treated)) | 193
Completed | 146
Not Completed | 47
Not completed — Adverse Event | 4
Not completed — Insufficient Effectiveness | 8
Not completed — Improved | 12
Not completed — Lost to Follow-up | 7
Not completed — Other than specified | 3
Not completed — No visit after the first visit | 13

BASELINE CHARACTERISTICS:
Population: Patients in safety set included patients ≥ 15 years old diagnosed with mild to moderate persistent bronchial asthma who are naive to Spiriva Respimat and received Spiriva Respimat for the first time for treatment of bronchial asthma on top of at least inhaled corticosteroid (ICS) treatment
Arm/Group | Spiriva Respimat Group
Number analyzed (Participants) | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suspected Adverse Drug Reactions (ADRs)
Description: Number of participants with suspected adverse drug reactions (ADRs) is presented.
  An Adverse Event (AE) was considered to be ADR if either the physician who reported the AE or the sponsor assessed its causal relationship as related.
Time Frame: From first drug administration until 30 days after last drug administration; up to 337 days
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Spiriva Respimat Group
Number analyzed (Participants) | 180
Participants | 5

2. Secondary Outcome: The Change From Baseline in Asthma Control Status at Week 12 Using Asthma Prevention and Management Guideline
Description: The change from baseline in asthma control status at week 12 using Asthma prevention and management guideline is presented.
  Well controlled is a better outcome compared to Insufficiently controlled and Poorly controlled outcomes.
  Abbreviations used:
  Baseline (BL), Week 12 (W12), Well-controlled (WC), Insufficiently controlled (IC), Poorly controlled (PC), Unknown (UNK), Missing (MIS); If a patient was well-controlled at baseline and maintained the state until Week 12, the effectiveness was assessed as "no change". If a patient insufficiently controlled or poorly controlled at baseline became well-controlled at Week 12, or if a patient was poorly controlled at baseline and became insufficiently controlled at Week 12, Spiriva Respimat was assessed as "effective" (or the patient assessed as a responder). If the disease condition did not improve in a patient at Week 12 from baseline, Spiriva Respimat was assessed as "ineffective" (or the patient assessed as a non-responder).
Time Frame: baseline and 12 weeks
Population: Effectiveness set that excluded patients who were not associated with effectiveness data available (pulmonary function test or laboratory values related to asthma control status) as defined at baseline and/or on treatment.
Measure: Number; unit: participants
Arm/Group | Spiriva Respimat Group
Number analyzed (Participants) | 159
participants
  BL- WC W12-WC | 9
  BL-WC W12-IC | 0
  BL-WC W12-PC | 0
  BL-WC W12-UNK | 0
  BL-WC W12-MIS | 0
  BL-IC W12-WC | 68
  BL-IC W12-IC | 39
  BL-IC W12-PC | 0
  BL-IC W12-UNK | 0
  BL-IC W12-MIS | 6
  BL-PC W12-WC | 11
  BL-PC W12-IC | 10
  BL-PC W12-PC | 6
  BL-PC W12-UNK | 0
  BL-PC W12-MIS | 0
  BL-UNK W12-WC | 3
  BL-UNK W12-IC | 1
  BL-UNK W12-PC | 0
  BL-UNK W12-UNK | 4
  BL-UNK W12-MIS | 1
  BL-MIS W12-WC | 0
  BL-MIS W12-IC | 1
  BL-MIS W12-PC | 0
  BL-MIS W12-UNK | 0
  BL-MIS W12-MIS | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration; up to 337 days
Description: The safety set (The safety set includes all patients registered in the study and received the treatment) was used for adverse event reporting. A total of 193 patients were registered and Case Report Forms (CRFs) were collected from 193 patients. The safety set includes 180 patients, excluding 13 patients who had no visit after the first visit.
Groups:
- Spiriva Respimat Group: Patients with mild to moderate persistent asthma treated with Spiriva® 1.25 microgram (μg) Respimat® 60 puffs and Spiriva® 2.5 μg Respimat® 60 puffs (hereinafter, Spiriva Respimat). Daily dose was inhalation of the spray of two puffs of Spiriva 2.5 μg Respimat (5 μg of tiotropium) and the spray of two puffs of Spiriva 1.25 μg Respimat (2.5 μg of tiotropium) in this noninterventional, observational study to collect new real world data (i.e., data under routine medical practice)
Arm/Group | Spiriva Respimat Group
All-Cause Mortality (participants affected / at risk) | 0/180
Serious Adverse Events (participants affected / at risk) | 1/180
Other Adverse Events (participants affected / at risk) | 0/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva Respimat Group (N=180)
Herpes zoster (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Patients were not randomized and there are no within-study data. Patients in the study may differ from the overall asthma-treated population, or from treated patients who did not choose to participate in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03188120/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03188120/SAP_001.pdf